CLINICAL TRIAL: NCT03438019
Title: Inspiratory Muscle Strength and Endurance Training in Veterans With COPD
Brief Title: Inspiratory Muscle Training in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Campos, Principal Investigator, Miami VA Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160788-1
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: Maximal Respiratory Pressures, Inspiratory Muscle Training, TIRE, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TIRE IMT (Experimental): The TIRE IMT group will receive a tablet with the TIRE software installed and a PrO2® device through which they will train. Training consists of six levels (A-F) with six inspirations at each level for a total of 36 breaths. Recovery times between breaths range from 40 to 5 seconds as the subject advances each level. TIRE data will be stored in the tablet for subsequent interrogation and data retrieval.
  Interventions: Device: PrO2
- Standard IMT group (Experimental): The Standard IMT group will receive a Threshold® Inspiratory Muscle Trainer. This device incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting to be set based on MIP values of each subject. Subjects will be instructed to perform up to 36 breaths daily. To compare with TIRE training, we will ask participants to perform this within a 30-minute session.
  Interventions: Device: Threshold Inspiratory Muscle Trainer
- Sham IMT group (Sham Comparator): The Sham IMT group will also receive a Threshold® device and undergo the exact protocol of group 2 but with minimal resistance applied (7 cm H2O, the lowest in the device).
  Interventions: Device: Threshold Inspiratory Muscle Trainer

INTERVENTIONS:
Device: PrO2 — The PrO2 device is linked to a tablet via Bluetooth and provides the user with a graphic representation of their inspiratory effort throughout all of inspiration and real-time biofeedback. This device incorporates a standard 2mm leak to avoid glottal closure during maximal inspiration. The PrO2 provides measures of MIP (cmH2O), SMIP (PTU) and ID (seconds).
  Other Names: TIRE
  Arms: TIRE IMT
Device: Threshold Inspiratory Muscle Trainer — The Threshold incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting to be set based on MIP values of each subject.
  Arms: Sham IMT group; Standard IMT group

SUMMARY:
This proposal aims at evaluating an inspiratory muscle training (IMT) method not previously tested in COPD called the Test of Incremental Respiratory Endurance (TIRE). As a training method, TIRE promises to provide further benefits over standard IMT because it allows the user to adjust training loads as progress is made, adjusts the training based on day-to-day variations commonly noted in COPD, and provides a graphic representation of the inspiratory effort throughout all inspiration with real-time biofeedback in order to "coach" the user in performing the exercises. The TIRE device can also be used as an assessment tool, not only to measure the commonly used measure of inspiratory muscle strength Maximal Inspiratory Pressure (MIP), but also measuring the MIP variation generated throughout a maximal sustained inspiration. In this way, TIRE integrates MIP over the inspiratory duration (ID), providing a novel derivative measure called the sustained maximal inspiratory pressure or SMIP, that is likely a better surrogate of inspiratory muscle performance in COPD based upon preliminary data. The main goal of this trial is to fully evaluate the utility of TIRE as an IMT method in veterans with COPD. The investigators hypothesize that as a stand-alone therapy, TIRE training is superior to standard IMT in improving inspiratory muscle strength and endurance and in improving COPD-related clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged > 40 years with a confirmed diagnosis of COPD by a pulmonologist (presence of risk factors and airflow obstruction) and evidence of inspiratory muscle weakness as defined by the latest American Thoracic Society / European Respiratory Society statement on respiratory muscle training.

Exclusion Criteria:

* Refusal to participate in the study, subjects actively undergoing pulmonary rehabilitation, inability to perform the required maneuvers (i.e. patients with cerebrovascular accident or tracheostomy), subjects not in their stable state (i.e. having an acute exacerbation or within 4 weeks of having one) or presence of important comorbidities that may confound the interpretation of TIRE measures (i.e. decompensated heart failure, diaphragmatic paralysis, prior lung surgery, active cancer treatment, etc.). There will be no involvement of vulnerable populations.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Sustained Maximal Inspiratory Pressure (SMIP) | Change from baseline to 8 weeks.
  SMIP is obtained from a maximal sustained inspiratory effort performed through the TIRE method using the PrO2 device. SMIP is documented in pressure time units (PTU) and represents the area under the curve generated from the start to the end of inspiration, from residual volume to total lung capacity.

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Change from baseline to 8 weeks.
  MIP is obtained from a maximal inspiratory effort from residual volume using the TIRE software and recorded in centimeters of water.
Inspiratory Duration (ID) | Change from baseline to 8 weeks.
  ID is obtained from a maximal and sustained inspiratory effort using the TIRE software and recorded in seconds.

OTHER OUTCOMES:
Six-minute Walk Test (6MWT) | Change from baseline to 8 weeks.
  Sub-maximal exercise test used to assess aerobic capacity and endurance. The best distance covered over a time of 6 minutes is recorded in metres.
St.George's Respiratory Questionnaire (SGRQ) | Change from baseline to 8 weeks.
  The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
Modified Medical Research Council (mMRC) Dyspnea Scale | Change from baseline to 8 weeks.
  This scale ranges from zero to four, with higher scores indicating a greater degree of breathlessness.
COPD Assessment Test (CAT) | Change from baseline to 8 weeks.
  This instrument that can quantify the impact of COPD on the patient's health. The CAT has a scoring range of 0-40. Higher scores denote a more severe impact of COPD.
Fat Free Mass Index (FFMI) | Change from baseline to 8 weeks.
  FFMI is calculated using the following formula: FFMI = (Lean Mass / 2.2) / ((Height in feet * 12.0) * 0.0254) squared. A person is said to be in the Average Norms of Muscle Mass Interpretation when his FFMI in pounds is between 18 and 19.
Short Performance Physical Battery (SPPB) | Change from baseline to 8 weeks.
  The SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. The scores range from 0 (worst performance) to 12 (best performance).

CONTACTS AND LOCATIONS:
Locations (1):
- Bruce W Carter VAMC, Miami, Florida, United States